CLINICAL TRIAL: NCT01278615
Title: A Single-Arm Phase II Clinical Trial With the Novel MEK Inhibitor AZD-6244 for the Treatment of MCT-1 Related Relapsed or Refractory Diffuse Large B-Cell Lymphoma
Brief Title: Selumetinib in Treating Patients With Relapsed or Refractory Diffuse Large B-cell Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Closed Prematurely.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-02558; NCI-2011-02558 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NU-10H03; CDR0000690641; 12-0110 (Other: University of Chicago Comprehensive Cancer Center); 8611 (Other: CTEP); N01CM00071 (NIH); N01CM62201 (NIH); P30CA014599 (NIH)
Record Dates: First submitted 2011-01-15; First posted 2011-01-19 (Estimated); Results first posted 2016-02-03 (Estimated); Last update posted 2016-02-03 (Estimated); Status verified 2014-07

CONDITIONS: Recurrent Adult Diffuse Large Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — AZD 6244

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (selumetinib) (Experimental): Patients receive selumetinib PO BID on days 1-28. Treatment repeats every 28 days for 8 courses in the absence of disease progression or unacceptable toxicity
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Selumetinib

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Selumetinib — Given PO
  Other Names: ARRY-142886; AZD6244; MEK Inhibitor AZD6244

SUMMARY:
This phase II clinical trial is studying how well selumetinib works in treating patients with relapsed or refractory diffuse large B-cell lymphoma. Selumetinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the overall response rate (combined complete remission [CR] and partial remission [PR]) of AZD6244 hyd-sulfate anti-MEK (selumetinib) therapy for patients with relapsed or refractory diffuse large B-cell lymphoma (DLBCL).

SECONDARY OBJECTIVES:

I. To evaluate the safety and tolerability of MEK inhibitor therapy. II. To determine the progression-free survival, time to treatment failure, duration of response, and overall survival with AZD6244 hyd-sulfate therapy.

III. To examine biomarkers through down-regulation of phosphorylated extracellular signal-related kinase (pERK) and several relevant target substrates (e.g., monocarboxylate transporter-1 [MCT-1], Menkes disease-associated protein [MNK], ELK, c-v-myc avian myelocytomatosis viral oncogene homolog [c-MYC], and hypoxia-inducible factor-1alpha [HIF-1a]) in peripheral blood studies.

OUTLINE: This is a multicenter study.

Patients receive selumetinib orally (PO) twice daily (BID) on days 1-28. Treatment repeats every 28 days for 8 courses in the absence of disease progression or unacceptable toxicity.

Patients undergo blood sample and tumor tissue collection at baseline and at day 15 of course 1 for biomarker studies.

After completion of study therapy, patients are followed up every 3 months for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care
* Relapsed or refractory diffuse large B-cell lymphoma (transformed large cell lymphomas are allowed to enroll)
* Patients must have received at least one previous therapeutic regimen, and no more than 6 previous therapeutic regimens
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2
* Life expectancy > 3 months
* No chemotherapy, radiation therapy, immunotherapy, or experimental anticancer therapy within 28 days before beginning study treatment
* Human immunodeficiency virus (HIV)-positive patients are eligible if: the cluster of differentiation (CD)4 count is > 400, have no acquired immune deficiency syndrome (AIDS)-defining illnesses (other than non-Hodgkin lymphoma [NHL]), and they are not taking combination antiretroviral therapy (cART) at the time of study entry that would interfere with cytochrome P450, family 3, subfamily A, polypeptide 4 (CYP4503A4)
* No other active infection
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control, or abstinence) prior to study entry, for the duration of study participation, and for 4 weeks after dosing with AZD6244 hyd-sulfate ceases; women of child-bearing potential must have a negative pregnancy test prior to entry; should a woman become pregnant or suspect she is pregnant while she or her partner participating in this study, the patient should inform her treating physician immediately; please note that the AZD6244 hyd-sulfate manufacturer recommends that adequate contraception for male patients should be used for 16 weeks post-last dose due to sperm life cycle
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated with AZD6244 hyd-sulfate
* Patients may have received prior autologous, but not prior allogeneic stem cell transplant; however, patients who are eligible for potentially curative treatment with bone marrow transplant should not be entered on this investigational trial, unless they refuse the transplant option (or are not eligible for transplantation)

Exclusion Criteria:

* Any prior exposure to mitogen-activated protein kinase kinase (MEK), Ras, or v-raf murine sarcoma 3611 viral oncogene homolog (Raf) inhibitors
* Patients with any active central nervous system (CNS) involvement by lymphoma are excluded
* Patients that are taking drugs that alter CYP450 3A4 (or cannot be changed to drugs that do not alter CYP450 3A4) are excluded
* Cardiac conditions as follows:

  * Uncontrolled hypertension (blood pressure [BP] >= 150/95 despite optimal therapy)
  * Heart failure New York Heart Association (NYHA) class II or above
  * Prior or current cardiomyopathy
  * Baseline left ventricular ejection fraction (LVEF) =< 50%
  * Atrial fibrillation with heart rate > 100 beats per minute (bpm)
  * Unstable ischemic heart disease (myocardial infarction [MI] within 6 months prior to starting treatment, or angina requiring use of nitrates more than once weekly)
  * Patients are excluded if there is corrected QT (QTc) interval > 450 msecs or other factors that increase the risk of QT prolongation or arrhythmic events (e.g., heart failure, hypokalemia, family history of long QT interval syndrome)
  * Patients are excluded if they are taking any drugs that may significantly prolong the QTc; these drugs are prohibited during the study; if the patient is taking one or more of these medications, they may enroll if all pertinent medications are stopped with the associated "wash out" periods
* Absolute neutrophil count (ANC) < 1.5 x 10^9/L (1500 per mm^3)
* Platelets < 100 x 10^9/L
* Hemoglobin (Hgb) < 8.0 g/dL
* Serum bilirubin >= 1.5 x upper limit of normal (ULN)
* Aspartate aminotransferase (AST/serum glutamic oxaloacetic transaminase [SGOT]) or alanine aminotransferase (ALT/serum glutamate pyruvate transaminase [SGPT]) >= 2.5 x ULN (>= 5 ULN in presence of liver metastases)
* There should be a minimum of a 1 month wash-out interval from another investigational product to AZD6244 hyd-sulfate dosing start plus recovery from side effects of investigational product
* There should be a minimum of a 1 month wash-out interval from the end of previous systemic treatment and radiotherapy
* Patients are excluded if there is a history of a serious medical or psychiatric illness likely to interfere with participation in this clinical study
* Patients may not have recent history of refractory nausea and vomiting, chronic gastrointestinal diseases (e.g., inflammatory bowel disease), or significant bowel resection that would preclude adequate absorption

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2010-12; Primary Completion 2014-02 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leo Gordon, Principal Investigator — Northwestern University
Locations (16):
- United States (16):
  - Northwestern University, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Southern Illinois University, Springfield, Illinois
  - Fort Wayne Medical Oncology and Hematology Inc-Parkview, Fort Wayne, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - University of Massachusetts Memorial Health Care, Worcester, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Saint John's Mercy Medical Center, St Louis, Missouri
  - Weill Medical College of Cornell University, New York, New York
  - M D Anderson Cancer Center, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Selumetinib)
Started | 16
Completed | 14
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Selumetinib)
Number analyzed (Participants) | 16
Age, Continuous [Median (Full Range); unit: years] | 70 [28.7 to 86.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 9

OUTCOME MEASURES:

1. Primary Outcome: Response Rate (Complete Response [CR] and Partial Response [PR]) in Patients Treated With Selumetinib
Description: Estimates of the response rate based on best response (CR and PR) with the exact two-sided 95% confidence intervals. Response for this lymphoma clinical study was measured utilizing "Non-Hodgkins Lymphoma Response Criteria". These criteria are based upon the criteria from the Revised Response Criteria for Malignant Lymphoma, (Cheson et al.), Journal of Clinical Oncology, 2007, Vol. 25:579-586.
Time Frame: Up to 3 years
Measure: Number (95% Confidence Interval); unit: percentage of response
Arm/Group | Treatment (Selumetinib)
Number analyzed (Participants) | 14
percentage of response | 0 [0 to 23]

2. Secondary Outcome: Duration of Response
Description: The Kaplan-Meier procedure will be used to characterize the duration of response. Median time-to-event and the corresponding two-sided 95% confidence intervals will be provided.
Time Frame: From the documented beginning of response (CR or PR) to the time of relapse, assessed up to 3 years
Population: Zero participants were analyzed due to no response.
Arm/Group | Treatment (Selumetinib)
Number analyzed (Participants) | 0

3. Secondary Outcome: Incidence of Adverse Events Graded Using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0
Description: Percentage of patients experiencing any grade 3 or higher adverse event at least possibly attributed to the study drug. (Additional adverse event reporting will appear in the AE outcomes module.)
Time Frame: Up to 3 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Selumetinib)
Number analyzed (Participants) | 16
percentage of participants | 37.5 [15.2 to 64.6]

4. Secondary Outcome: Overall Survival
Description: The Kaplan-Meier procedure will be used to characterize the survivorship function. Median time-to-death and the corresponding two-sided 95% confidence intervals will be provided.
Time Frame: Date of study entry to the date of death, assessed up to 3 years
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Treatment (Selumetinib)
Number analyzed (Participants) | 14
days | 129 [58 to 134]

5. Secondary Outcome: Progression-free Survival
Description: The Kaplan-Meier procedure will be used to characterize the survivorship function. Median time-to-event and the corresponding two-sided 95% confidence intervals will be provided.
Time Frame: Time from entry onto study until lymphoma progression or death from any cause, assessed up to 3 years
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Treatment (Selumetinib)
Number analyzed (Participants) | 14
days | 34 [14 to 73]

6. Secondary Outcome: Time to Treatment Failure
Description: as for outcome 5
Time Frame: Time from study entry to treatment failure, defined as lymphoma progression or withdrawal from treatment due to adverse events, assessed up to 3 years. Patients who die without progression while still on therapy will be censored as of the time of death.
Measure: Mean (95% Confidence Interval); unit: days
Arm/Group | Treatment (Selumetinib)
Number analyzed (Participants) | 14
days | 34 [14 to 73]

7. Primary Outcome: Disease Control Rate (Complete Response [CR], Partial Response [PR], and Stable Disease [SD]) in Patients Treated With Selumetinib
Description: Estimates of the disease control rate with the exact two-sided 95% confidence intervals. Response was measured utilizing "Non-Hodgkins Lymphoma Response Criteria". These criteria are based upon the criteria from the Revised Response Criteria for Malignant Lymphoma, (Cheson et al.), Journal of Clinical Oncology, 2007, Vol. 25:579-586. Using these criteria, 'disease control rate' encompassed patients who had either a CR, PR, and SD.
Time Frame: Up to 3 years
Measure: Number (95% Confidence Interval); unit: percentage of disease control
Arm/Group | Treatment (Selumetinib)
Number analyzed (Participants) | 14
percentage of disease control | 14.3 [1.8 to 42.8]

ADVERSE EVENTS:
Arm/Group | Treatment (Selumetinib)
Serious Adverse Events (participants affected / at risk) | 7/16
Other Adverse Events (participants affected / at risk) | 11/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Selumetinib) (N=16)
Anemia (Blood and lymphatic system disorders) | 1
Atrioventricular block complete (Cardiac disorders) | 1
Left ventricular systolic dysfunction (Cardiac disorders) | 1
Colonic obstruction (Gastrointestinal disorders) | 1
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1
Pancreatic necrosis (Gastrointestinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1
Death NOS (General disorders) | 1
Hypothermia (General disorders) | 1
Pain (General disorders) | 1
Skin infection (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 1
Injury to kidney (Injury, poisoning and procedural complications) | 2
Lymphocyte count decreased (Investigations) | 1
Neutrophil count decreased (Investigations) | 2
White blood cell decreased (Investigations) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Confusion (Psychiatric disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Hypotension (Vascular disorders) | 1
Thromboembolic event (Vascular disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Selumetinib) (N=16)
Anemia (Blood and lymphatic system disorders) | 7
Blurred vision (Eye disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 5
Dry mouth (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 1
Edema face (General disorders) | 2
Edema limbs (General disorders) | 3
Fatigue (General disorders) | 7
Fever (General disorders) | 2
Hypothermia (General disorders) | 1
Catheter related infection (Infections and infestations) | 1
Alanine aminotransferase increased (Investigations) | 3
Alkaline phosphatase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 7
Blood bilirubin increased (Investigations) | 1
Creatinine increased (Investigations) | 4
Electrocardiogram QT corrected interval prolonged (Investigations) | 1
Lymphocyte count decreased (Investigations) | 3
Neutrophil count decreased (Investigations) | 2
Platelet count decreased (Investigations) | 4
Weight gain (Investigations) | 1
White blood cell decreased (Investigations) | 3
Anorexia (Metabolism and nutrition disorders) | 4
Hypercalcemia (Metabolism and nutrition disorders) | 2
Hyperglycemia (Metabolism and nutrition disorders) | 6
Hypernatremia (Metabolism and nutrition disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 4
Hypocalcemia (Metabolism and nutrition disorders) | 4
Hypokalemia (Metabolism and nutrition disorders) | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 3
Metabolism and nutrition disorders Anorexia (Metabolism and nutrition disorders) | 4
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 1
Oral dysesthesia (Nervous system disorders) | 1
Paresthesia (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
Confusion (Psychiatric disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
Dry skin (Skin and subcutaneous tissue disorders) | 3
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 1
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1
Hypotension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less